CLINICAL TRIAL: NCT06621381
Title: A Single Group Evaluation of Concentrated Exposure and Response Prevention for Children With Obsessive-compulsive Disorder
Brief Title: Concentrated Exposure and Response Prevention for Children With Obsessive-compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Vendela Zetterqvist, Associate professor, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-07331-01
Record Dates: First submitted 2024-09-09; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-compulsive disorder; Exposure; Response prevention; Pediatric; Cognitive Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concentrated exposure and response prevention (Experimental): The intervention consists of: Psychoducation for the patients (1 session, 2-3h in group format), psychoeducation for the legal guardians (1 session, 3h in group format), exposure and response prevention (3-4 sessions, 9-12h over the course of one week, individual format), group reunions for sharing experiences, motivational work and relapse prevention ( 2 sessions, 3h)
  Interventions: Behavioral: Concentrated exposure and response prevention

INTERVENTIONS:
Behavioral: Concentrated exposure and response prevention — The intervention consists of: Psychoducation for the patients (1 session, 2-3h in group format), psychoeducation for the legal guardians (1 session, 3h in group format), exposure and response prevention (3-4 sessions, 9-12h over the course of one week, individual format), group reunions for sharing experiences, motivational work and relapse prevention ( 2 sessions, 3h)
  Other Names: cognitive behavioral therapy

SUMMARY:
The goal of this clinical trial is to evaluate the preliminary outcomes of concentrated exposure and response prevention for children with obsessive-compulsive disorder (OCD) in regular clinical practice. It is a non-randomised open label evaluation where children 6-12 years with OCD who are patients at the Child and Adolescent Psychiatry (CAP) at Uppsala University Hospital will be rectruited together with their legal guardians. The treatment will be delivered by trained therapists in regular outpatient care.

The main question the study aims to answer is:

What are the preliminary treatment effects of concentrated exposure and response prevention with regards to OCD-symptoms, functional impact, family accomodation and clinician ratings of severity and improvement?

Participants will receive psychoeducation (in group format) and exposure and response prevention (9-12h concentrated to one week, individual format).

Outcomes will be measured on structured interviews, clinician ratings, and validated questionnaires pre-treatment, post-treatment and at a six month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The patient fulfills the diagnostic criteria of obsessive-compulsive disorder
* The patient and the legal guardians have said yes to receiving the concentrated exposure with response prevention - treatment

Exclusion Criteria:

* The patient/legal guardians are unable to communicate in Swedish

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2029-12-14 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Childrens Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) | pre-intervention; one week after the intervention; six months after the intervention
  The Childrens Yale-Brown Obsessive-Compulsive Scale is a semi-structured interview made up of 10 items rated on a 5-point Likert scale evaluating the severity of Obsessions and Compulsions across five dimensions; Frequency, Interference, Distress, Resistance, and Control, during the previous week and up to the time of interview. The total score varies between 0 and 40. Higher scores indicate higher severity of Obsessions and Compulsions.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | pre-intervention; one week after the intervention; six months after the intervention
  The Clinical Global Impression is a brief, stand-alone assessment of the clinicians view of the patients global functioning prior to and after initiating treatment. It comprises two one-item measures evaluating (a) severity of psychopathology from 1 to 7 where a higher score indicates a higher severity, and (b) change from the initiation of treatment from 1 to 7, where a lower score indicates more improvement (1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse)
Dimensional Obsessive-Compulsive Scale - Child Version (DOCS-CV) | pre-intervention; one week after the intervention; six months after the intervention
  The Dimensional Obsessive-Compulsive Scale - Child Version is a 20-item self-report instrument that assesses the severity of Obsessive-Compulsive Disorder (OCD) symptoms along four empirically supported theme-based dimensions: (a) contamination, (b) responsibility for harm and mistakes, (c) incompleteness/symmetry, and (d) unacceptable (taboo) thoughts.over the preceding one month. The scale is developed for children and adolescents aged 7 to 17 years. Within each subscale, the five item scores are summed to produce a subscale score (range = 0-20). The four subscale scores can be summed to produce an overall DOCS total score (range = 0-80). Higher score indicate higher severity of Obsessive-Compulsive Disorder.
The Obsessive Compulsive Inventory-Child Version (OCI-CV) | pre-intervention; one week after the intervention; six months after the intervention
  A 21-item self-report measure that assesses obsessive compulsive symptoms in children and adolescents aged 7 to 17 years over the preceding one month. It is a Likert-type rating scale, scored 0 to 2 (where 0 = never, 1 = sometimes and 2 = always). The total score varies between 0 and 42 where higher scores indicate more symptoms.
Dimensional Obsessive-Compulsive Scale - Parent Version (DOCS-PV) | pre-intervention; one week after the intervention; six months after the intervention
  The Dimensional Obsessive-Compulsive Scale - Parent Version is a 20-item self-report instrument that assesses the severity of Obsessive-Compulsive Disorder (OCD) symptoms along four empirically supported theme-based dimensions: (a) contamination, (b) responsibility for harm and mistakes, (c) incompleteness/symmetry, and (d) unacceptable (taboo) thoughts.over the preceding one month. The scale is developed for parents or legal guardians to children and adolescents aged 7 to 17 years. Within each subscale, the five item scores are summed to produce a subscale score (range = 0-20). The four subscale scores can be summed to produce an overall DOCS total score (range = 0-80). Higher score indicate higher severity of Obsessive-Compulsive Disorder.
The Family Accommodation Scale for Obsessive Compulsive Disorder - Self-Rated Version (FAS-SR) | pre-intervention; one week after the intervention; six months after the intervention
  Parental assessment that aims to measure family members participation in or facilitation of rituals and/or avoidance in obsessive-compulsive disorder.
  The first section consists of a symptom checklist for Obsessive Compulsive Disorder. The second section contains 19 items that examine the frequency of accommodating behaviors carried out by the relative. Each item is rated on a 5-point scale (0 = none/never, 4 = every day). The total score varies between 0 and 76 points. Higher scores indicate more family accommodation.

CONTACTS AND LOCATIONS:
Overall Officials: Vendela Zetterqvist, Ph D, Associate Professor, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Region Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to restrictions in Swedish legislation